CLINICAL TRIAL: NCT02891902
Title: Impact of Dedicated Hygienist Staff on the Occurrence of Intensive Care Unit -Aquired Bloodstream Infections
Acronym: BacterHy
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_3682
Record Dates: First submitted 2016-08-31; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-08

CONDITIONS: Intensive Care Unit -Aquired Bloodstream Infections.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: hygienist response — The daily presence of a public health nurse in the intensive care unit would implement such a strategy for prevention of infections and reduce the incidence of bloodstream infections acquired in intensive care.

SUMMARY:
The purpose of this study is to evaluate in a multicentric cluster randomized study the effect of the presence of dedicated nurses for training of ICU staff in preventing nosocomial infections. The rate of bloodstream infections per 100 admitted patients is used as the main endpoint. A sample of 4000 included patients in the 6 participating ICU is included with the objective to show a reduction of one third of the rate of ICU-acquired bloodstream infections. The study is currently at the end of the recrutimeent phase.

DETAILED DESCRIPTION:
15% of patients admitted to intensive care have an infection acquired in the service, including bacteremia is a serious form. Compliance with hygiene measures and recommendations in the use of invasive devices can reduce the incidence. The advantage of simple recommendations type "bundle" could, however, be insufficient because not associated with training and monitoring compliance with the recommendations. The aim of this study is to show that the daily intervention of a public health nurse on the basis of a half full-time equivalent, allows these actions and therefore a reduction in the bloodstream of the attack rate acquired in the ICU compared dissemination of simple recommendations.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to reanimation department

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients admitted to reanimation department
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
rate of first ICU acquired bloodstream infection for 100 admitted patients | 2 months
  Collection of blood cultures

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hopital Nord Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No